CLINICAL TRIAL: NCT05480852
Title: Clinical Performance of BIS-GMA Free Dental Resin Composite as Posterior Restoration: a Randomized Clinical Trial
Brief Title: Clinical Performance of BIS-GMA Free Dental Resin Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Reda Mohamed, Assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Faculty of Dentistry
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Therapeutics
Keywords: Bis-GMA free dental resin composite; Bis-GMA containing dental resin composite; Clinical performance; Modified US Public Health Service Clinical Criteria (USPHS)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bis-GMA Free dental resin composite (Experimental): Restorative Materials
  Interventions: Other: Bis-GMA Free dental resin composite
- Bis-GMA containing dental resin composite (Active Comparator): Restorative Materials
  Interventions: Other: Bis-GMA Free dental resin composite

INTERVENTIONS:
Other: Bis-GMA Free dental resin composite — Restorative Material

SUMMARY:
Resin composites were introduced for restoring defective teeth commercially in the mid- 1960s as an alternative to acrylic resin and silicate cements. As one of the most signiﬁcant contributions to dentistry, dental resin composites usually have three components as organic resin matrix, photo initiator system, and coupling agent treated inorganic ﬁllers.

At present, the most commonly used organic resin matrix for dental resin composites are based on di-methacrrylates such as 2.2- bis [p-(2- hydroxy-3- methacryloxypropoxy) penylene] propane (Bis-GMA), ethoxylated bisGMA, 1,6-bis(2-methacryloyoxy-ethoxycarbonyl-amino)-2,4,4tri-methyl-hexane (UDMA) and triethyleneglycoldimethacrylate (TEGDMA).

The application of Bis-GMA has been doubted since it was reported to have estrogenic activity in a cell culture assay.Though later studies have showed that Bis-GMA does not hydrolyse into the estrogenic substance BPA, BPA has still been detected to be release out of several commercial Bis-GMA-based dental restorative materials. Although there is a lack of studies analysing the association between BPA exposure from dental materials and its adverse effects on human health, there is a need to develop newer BPA-free resin composites to minimize human exposure to this compound. Accordingly, the objective of this study was to evaluate the performance of BIS- GMA- free composite as a photopolymerizable posterior dental composite restoration.

DETAILED DESCRIPTION:
Hypothesis: The null hypothesis is that there is no difference in using the new BIS- GMA- free composite.

Aim of the study: This clinical trial was conducted to compare the clinical performance of the new BIS- GMA- free composite versus BIS-GMA- containing composite in the management of carious lesion in adult patients over 9 months. The two types of composites will be evaluated using USPHS criteria for:

* Retention (R).
* Contact (C).
* Color match (CM).
* Marginal adaptation (MA).
* Marginal discoloration (MD).
* Anatomic form (AF).
* Secondary caries (SC).
* Surface texture (ST).
* Gingival inflammation (GI).
* Post-operative sensitivity (POS).
* Patient complaints (PC).
* Patient satisfaction (PS).
* The evaluation done by three calibrated operators.

The study was conducted in Operative Dentistry Department, Faculty of Dentistry, Menia University.

The researcher was bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients, explaining, and performing the procedures to them.

- Intervention:

BIS- GMA- free composite material:

Tooth preparation and restoration was carried out using magnifying loops. All cavities were restored using composite resin. cavities, including the dentin, were acid etched for 30 s, rinsed thoroughly for 15 s, bonded with universal adhesive and light cured for 10 s prior to placing the filling material.

Restorations were light cured for 20 s, check the occlusion, finished with diamond burs and polished with Kenda hybrid composite pre- and super-polishers (Kenda, Vaduz, Liechtenstein).

- Comparator:

BIS- GMA- containing composite material:

The same methodology of the intervention BIS-GMA- free composite material If the patient showed any complications during our clinical trial toward either the intervention (BIS- GMA- free composite) or the comparator (BIS-GMA containing composite material), the trial will be stopped at once and all the needed management against any complications will be done.

ELIGIBILITY:
Inclusion Criteria:

* Have been from 20 to 45 years of age.
* Have at least two molars supported permanent dentition free of any clinically significant occlusal interference who required class I or class II restoration and fulfilled the inclusion criteria, will informed about the study and will give a patient information leaflet (PIL) describing their potential involvement.
* The two studied materials restorations should be used in approximately the same sized lesions or within the same extension.
* The patient will be reimbursed for attending for the clinical evaluation(s) of their restorations.
* Be a regular dental attender who agree to return for assessments.

Exclusion Criteria:

* There was a history of any adverse reaction to clinical materials of the type to be used in the study.
* There was evidence of occlusal parafunction and/or pathological tooth wear.
* patients whose history revealed parafunctional habits or use of medications that potentially could cause hyposalivation.
* They are pregnant or have medical and/or dental histories which could possibly complicate their attendance for the assessment of the restorations and/ or influence the behavior and performance of the restorations in the clinical service.
* They were irregular dental attenders.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of BIS- GMA- free composite as a photopolymerizable posterior dental composite restoration versus BIS-GMA containing composite. | 9 months
  This clinical trial conducted to compare the clinical performance of the new BIS- GMA- free composite versus BIS-GMA- containing composite in the management of carious lesion in adult patients over 9 months. The two types of composites will be evaluated using USPHS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Reda, Phd, Principal Investigator — Faculty of Dentistry, Minia University
Locations (1):
- Sara Ahmed Reda Mohamed, Minya, Egypt

REFERENCES:
- [Derived] Reda SA, Hussein YF, Riad M. The impact of Bis-GMA free and Bis-GMA containing resin composite as posterior restoration on marginal integrity: a randomized controlled clinical trial. BMC Oral Health. 2023 Dec 19;23(1):1022. doi: 10.1186/s12903-023-03759-5. PMID 38114979